CLINICAL TRIAL: NCT06586580
Title: Le Traitement Par Lenvatinib + Anti-PD1 Du Mélanome Métastatique
Brief Title: Treatment of Metastatic Melanoma with Lenvatinib + Anti-PD1
Acronym: LENVAMEL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/757
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Metastatic melanoma: Metastatic melanoma refractory to immunotherapy

SUMMARY:
The hypothesis is that treatment with Lenvatinib + Pembrolizumab is less effective in real life than in clinical trials. In fact, an objective response rate < 20% and a worse tolerability of the treatment in real life with ≥50% of severe toxicities are expected.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic melanoma (stage III non operable or stage IV according to American Joint Committee on Cancer staging rules) refractory to immunotherapy (≥ 2nd treatment line after minimum a failure of immunotherapy)

Exclusion Criteria:

* Uveal melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic melanoma (stage III non operable or stage IV according to AJCC)
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Month 18

SECONDARY OUTCOMES:
Progression-free survival | Month 18
Overall survival | Month 18
Frequencies of severe toxicities leading to treatment interruption | Month 18
  According to Common Terminology Criteria for Adverse Events [CTACE] V5, grade III and IV

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No